CLINICAL TRIAL: NCT02071927
Title: A Phase 1 Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Escalating Oral Doses of the Glutaminase Inhibitor CB-839 in Patients With Relapsed and/or Treatment-Refractory Leukemia
Brief Title: Study of the Glutaminase Inhibitor CB-839 in Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-003
Record Dates: First submitted 2014-02-14; First posted 2014-02-26 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukemia (ALL)
Keywords: leukemia; glutaminase; glutamine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — CB-839; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CB-839 (Experimental): CB-839 administered as oral capsules two (BID) or three times daily (TID) in 21-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839
- CB-Aza (Experimental): CB-839 administered as oral capsules twice daily (BID) in combination with azacitidine in 28-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839; Drug: CB-Aza

INTERVENTIONS:
Drug: CB-839 — Single-agent CB-839
  Other Names: Glutaminase inhibitor
Drug: CB-Aza — CB-839 in combination with standard dose azacitidine
  Other Names: combo CB-839 and azacitidine
  Arms: CB-Aza

SUMMARY:
Many tumor cells, in contrast to normal cells, have been shown to require the amino acid glutamine to produce energy for growth and survival. To exploit the dependence of tumors on glutamine, CB-839, a potent and selective inhibitor of the first enzyme in glutamine utilization, glutaminase, will be tested in this Phase 1 study in patients with leukemia.

This study is an open-label Phase 1 evaluation of CB-839 in subjects with leukemia. Part 1 is a dose escalation study to identify the recommended Phase 2 dose as a single agent and in combination with azacitidine. Patients enrolled into Part 2 will be treated with the recommended Phase 2 dose. As an extension of Part 2, patients with relapsed/ refractory or newly diagnosed AML will be treated with CB-839 in combination with azacitidine.

All patients will be assessed for safety, pharmacokinetics (plasma concentration of drug), pharmacodynamics (inhibition of glutaminase), biomarkers (biochemical markers that may predict responsiveness in later studies), and tumor response.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of AML or ALL, relapsed or refractory after at least 1 prior treatment regimen. Newly-diagnosed patients ≥ 60 years old who have refused or are considered unfit for standard chemotherapy regimens or stem cell transplantation are also eligible.
* Patients must have no available approved therapies that confer clinical benefit
* All patients must have bone marrow involvement of their tumor, with documented blast percentage of > 5%.
* Peripheral blood blast count must be ≤ 30,000 cells/µL.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate hepatic, renal, and cardiac function

Exclusion Criteria

* Any other current malignancy
* Patients with acute promyelocytic leukemia (APL)
* Treatment with an unapproved, investigational agent within 21 days of the first dose of study drug
* Allogeneic hematopoietic stem cell transplant or Donor Lymphocyte Infusion within 90 days prior to to the first dose of study drug
* Active GVHD
* Unable to receive medications by mouth
* Major surgery within 28 days before Cycle 1 Day 1
* Uncontrolled, active infection; patients who are known to have HIV infection/ seropositivity, Hepatitis A, B, or C, or CMV reactivation
* Significant neurotoxicity/neuropathy (Grade 3 or higher) within 14 days prior to Day 1
* Refractory nausea and vomiting or other situation that may preclude adequate absorption
* Conditions that could interfere with treatment and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CB-839: Incidence of adverse events | Every 21 days from study start until disease progression or unacceptable toxicity, assessed an expected average of 6 months

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the Curve (AUC) of CB-839 concentration in blood | Study Days 1, 15, and 22
Pharmacodynamics: % inhibition of glutaminase in blood | Study Days 1 and 15
Clinical Activity: % of Tumor Cells in Bone Marrow | Every 21 days from study start, assessed for an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith W Orford, MD, PhD, Study Director — Calithera Biosciences
Locations (5):
- United States (5):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179